CLINICAL TRIAL: NCT02955095
Title: Usability and Pilot Testing - Intervention for Smoking Cessation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn due to lack of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01288
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Current cigarette smoker (Experimental)
  Interventions: Device: Quit Smoking Phone Application

INTERVENTIONS:
Device: Quit Smoking Phone Application — The app will be downloaded on participants' phones, and used by the participant for 30 days to make a quit attempt. Participants will be encouraged to use the app every day and to utilize all of its features, including features such as setting a quit date, taking the assessment section, and entering cigarette use and reasons for cravings

SUMMARY:
The purpose of the usability and pilot testing for the project "Developing a Bi-national Buddy Intervention for Smoking Cessation and Cultural Education" is to better understand how users interact with the smoking cessation app, and to improve the product based on the results. In pilot testing the smoking cessation app the investigators will examine the feasibility of our approach. The usability testing portion of the study is intended primarily to improve on the design of the smoking cessation app, and will: gather quantitative data on participant's performance, identify usability problems, and determine user satisfaction with the app. The pilot testing portion of the study will evaluate the feasibility, time, cost and statistical variability in an attempt to predict an appropriate sample size and improve upon the study design prior to performance of a full-scale research study.

Objective 1:To collect quantitative data on participant's performance while using the app for smoking cessation.

Objective 2:To identify problems with usability of the smoking cessation buddy app.

Objective 3:To assess user satisfaction with the smoking cessation buddy app. Objective 4:To improve upon the design of the smoking cessation buddy app Objective 5:To assess the feasibility, time, cost, and statistical variability for a full-scale implementation of this study with the intervention group.

DETAILED DESCRIPTION:
Tobacco use cessation among youth is not adequately addressed in the US and Russia. The proposed intervention utilizes an innovative evidence-based approach while addressing the shortcomings of prior individual intervention components. In this project, investigators seek to refine a smoking cessation app by conducting two rounds of usability testing followed by a pilot test of the final app, to access usability problems, user satisfaction, and user-friendliness. This data will be collected in a de-identified and confidential manner, and will then be analyzed and used to refine the final app that will later be used.

ELIGIBILITY:
Inclusion Criteria:

* Current student
* Current cigarette smoker (smoked in past 30 days)
* speak English
* Own a smartphone
* Has some interest in quitting smoking.

Exclusion Criteria:

* Not meeting inclusion criteria.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Cigarettes smoked per day | 30 Days
How many times the app is accessed, | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sherman, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States